CLINICAL TRIAL: NCT00126906
Title: Intermittent Preventive Treatment With Sulfadoxine/Pyrimethamine During Pregnancy Among HIV-Positive and HIV-Negative Women: 2-Dose Versus Monthly - Malawi
Brief Title: Prevention of Malaria During Pregnancy Using Intermittent Preventive Treatment With Sulfadoxine-Pyrimethamine: Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Health and Population, Malawi (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: CDC-NCID-3429
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2005-08-23 (Estimated); Status verified 2005-08

CONDITIONS: Malaria, Falciparum; HIV Infections
Keywords: Malaria; Pregnancy; HIV
MeSH Terms: conditions — Malaria, Falciparum; HIV Infections; Malaria | interventions — Pyrimethamine; Sulfadoxine

INTERVENTIONS:
Drug: Monthly sulfadoxine/pyrimethamine
Drug: 2-dose sulfadoxine/pyrimethamine

SUMMARY:
In Malawi, the standard of care to prevent malaria during pregnancy at the time of the study was a two dose sulfadoxine-pyrimethamine intermittent protective treatment (SP IPT) regimen administered in the second and third trimester of pregnancy. In this investigation, this two dose strategy was compared to a monthly SP regimen. The objective for the study was to determine the efficacy of the different regimens for HIV positive and HIV negative women in the prevention of placental malaria.

DETAILED DESCRIPTION:
In this protocol the researchers wish to elaborate prior investigations on factors which may affect prevalence and malarial parasite density in pregnant women in Malawi. Primarily, this investigation will evaluate the efficacy of the current Malawian national policy, sulfadoxine-pyrimethamine (SP) 2-dose intermittent protective treatment (IPT) strategy, and compare it to a monthly SP strategy for use in preventing malaria during pregnancy. Previous investigations in Malawi have demonstrated that: prevention of malaria during pregnancy is most important during the first and second pregnancies, particularly during the rainy season when malaria transmission is highest; and an efficacious antimalarial regimen which clears parasitemia and placental infection will result in a reduction in the incidence of low birth weight, the single greatest risk factor for neonatal and early infant mortality. There appears to be an interaction between HIV infection and placental malaria, with HIV-positive pregnant women having higher prevalences and densities of peripheral and placental parasitemia compared with HIV-negative pregnant women. This finding requires closer examination, in light of the high prevalence and incidence of HIV infection in Malawi and other African countries. Previously in Malawi, a 2-dose IPT regimen of SP administered during the second and third trimester of pregnancy was effective at clearing placental malaria infection at delivery More recent studies in both Malawi and Kenya show that 2 doses may not be adequate in clearing placental parasitemia especially in women who are HIV infected. In the Kenya study, HIV-positive women required 3 doses of SP (that were delivered in a monthly dosing scheme) to achieve similar reductions in placental parasitemia that were seen in HIV-negative women at 2 doses. There remains a need to identify the optimal dosing schedule for an intermittent treatment regimen; the Kenya findings need to be confirmed before decisions are made on national and global levels. This is especially important given the possibility of increasing SP resistance in Malawi. The question of HIV infection and its role in malaria during pregnancy, both in terms of impact on regimen effectiveness and on the incidence of adverse sulfa reactions needs to be examined. This study proposes to determine the efficacy of the current regimen of 2-dose SP intermittent protective treatment (IPT) and to compare it to monthly SP dosing in clearing placental parasitemia at delivery in Machinga district in Malawi where there is a high level of malaria transmission and an HIV seropositivity rate of nearly 20% in reproductive age woman. This study will also explore the effect of HIV seropositivity on the safety and efficacy of intermittent preventive treatment during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* First or second pregnancy
* Greater than 16 weeks gestation
* Less than 28 weeks gestation
* Consent for HIV testing

Exclusion Criteria:

* Less than 15 years old

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700
Dates: Start 2002-10; Study Completion 2005-03

PRIMARY OUTCOMES:
Placental malaria parasitemia rates measured at time of delivery, stratified by HIV status

SECONDARY OUTCOMES:
Proportion of newborns with low birth weight, stratified by HIV status
Proportion of women with third trimester anemia, stratified by HIV status
Proportion of pregnancies that suffer fetal loss, stratified by HIV status

CONTACTS AND LOCATIONS:
Overall Officials: Scott J Filler, MD, DTM&H, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Machinga District Hospital, Liwonde, Malawi

REFERENCES:
- [Background] Parise ME, Ayisi JG, Nahlen BL, Schultz LJ, Roberts JM, Misore A, Muga R, Oloo AJ, Steketee RW. Efficacy of sulfadoxine-pyrimethamine for prevention of placental malaria in an area of Kenya with a high prevalence of malaria and human immunodeficiency virus infection. Am J Trop Med Hyg. 1998 Nov;59(5):813-22. doi: 10.4269/ajtmh.1998.59.813. PMID 9840604
- [Derived] Pons-Duran C, Wassenaar MJ, Yovo KE, Marin-Carballo C, Briand V, Gonzalez R. Intermittent preventive treatment regimens for malaria in HIV-positive pregnant women. Cochrane Database Syst Rev. 2024 Sep 26;9(9):CD006689. doi: 10.1002/14651858.CD006689.pub3. PMID 39324693
- [Derived] Filler SJ, Kazembe P, Thigpen M, Macheso A, Parise ME, Newman RD, Steketee RW, Hamel M. Randomized trial of 2-dose versus monthly sulfadoxine-pyrimethamine intermittent preventive treatment for malaria in HIV-positive and HIV-negative pregnant women in Malawi. J Infect Dis. 2006 Aug 1;194(3):286-93. doi: 10.1086/505080. Epub 2006 Jun 20. PMID 16826475